CLINICAL TRIAL: NCT02024269
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells Injected Intravitreal in Dry Macular Degeneration
Brief Title: Study to Assess the Safety and Effects of Cells Injected Intravitreal in Dry Macular Degeneration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Bioheart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADI-US-AMD-001
Record Dates: First submitted 2013-12-17; First posted 2013-12-31 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Dry Macular Degeneration
Keywords: macular degeneration; stem cells; adipose stem cells
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

ARMS (1):
- Adipose Stem Cells (Experimental)
  Interventions: Biological: Adipose Derived Stem Cells

INTERVENTIONS:
Biological: Adipose Derived Stem Cells

SUMMARY:
This will be an open-label, non-randomized multi-center study of adipose stem cell (ASC) implantation. ASCs will be derived from the patient's adipose or fat. Liposuction using local anesthesia and syringe collection will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells. The cells will be delivered via needle injection into the eye.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between Age 50 and 90 years
* Patients with dry AMD
* Visual acuity in the study eye <20200 (equal to or worse than 20/200)

Exclusion Criteria:

* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Inability to undergo syringe liposuction procedure or have any medical problems that contraindicate the procedure.
* Life expectancy < 6 months due to concomitant illnesses.
* Vitrectomized eyes
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease. . If patients have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis, an expert will be consulted as to patient eligibility based on the patient's infectious status
* Any illness which might affect a patient's survival over the follow-up period
* Any illness which, in the Investigator's judgement, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Patients with severe coagulation disorders
* Systolic blood pressure (supine) ≤90 mmHg;
* Resting heart rate > 100 bpm;
* Active clinical infection being treated by antibiotics within one week of enrollment.
* Cerebrovascular accident within 6 months prior to study entry
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* Severe COPD or severe asthma that would contraindicate surgery
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last two years.
* Unwilling and/or not able to give written informed consent.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
frequency and nature of adverse events | 6 months
Visual Field analysis (10-2) | 6 months
  Visual field testing can be performed clinically by keeping the subject's gaze fixed while presenting objects at various places within their visual field.
Visual Acuity Measurements | 6 months
  Visual acuity is a measure of the spatial resolution of the visual processing system. VA is tested by requiring the person whose vision is being tested to identify so-called optotypes - stylized letters, Landolt rings or other patterns - on a chart from a set viewing distance.

SECONDARY OUTCOMES:
Intraocular pressure | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bioheart, Sunrise, Florida, United States